CLINICAL TRIAL: NCT07070167
Title: Point-of-Care Ultrasonography for Assessing Lung Aeration and Pulmonary Vascular Resistance Dynamics After Surfactant Administration in Neonates With Respiratory Distress Syndrome
Brief Title: Bedside Ultrasound to Monitor Lung Function and Blood Flow in Newborns Treated With Surfactant
Acronym: ULISSES
Status: Not yet recruiting | Type: Observational
Sponsor: Chiesi Poland Sp. z o.o. (Industry)
Collaborators: Polish Ultrasound Society, Neonatal Section (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHI-PL-CUR-05
Record Dates: First submitted 2025-07-04; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Lung Ultrasound; Respiratory Distress Syndrome, Newborn
Keywords: surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Intratracheal administration of surfactant — Intratracheal administration of pulmonary surfactant with any of the approved methods: (a) via endotracheal tube in a mechanically-ventilated infant, (b) with the INSURE method (intubation-surfactant-extubation), or (c) with LISA method (through a thin catheter inserted intratracheally in a spontaneously breathing infant, supported with CPAP)

SUMMARY:
The ULISSES study looks at how doctors use bedside ultrasound to help treat premature babies with breathing problems caused by Respiratory Distress Syndrome (RDS). It focuses on whether doctors decide to give a medicine called surfactant based on oxygen levels alone or if they also use lung ultrasound images to guide their decision.

Around 200 babies will take part in the study in hospitals across Poland. Doctors will do ultrasound scans of the babies' lungs before and after surfactant is given. In some hospitals, heart and lung blood flow will also be checked to look for signs of high blood pressure in the lungs.

The study will see if both lungs improve equally after treatment or if one side stays worse, and whether this affects how much breathing support the baby needs. The results may help doctors improve how and when they give surfactant, leading to better care for newborns with RDS.

DETAILED DESCRIPTION:
The ULISSES study (Point-of-Care Ultrasonography for Assessing Lung Aeration and Pulmonary Vascular Resistance Dynamics After Surfactant Administration in Neonates With Respiratory Distress Syndrome) is a prospective, multicenter, non-interventional (observational) study involving approximately 200 preterm neonates across 10-12 tertiary-level neonatal intensive care units (NICUs) in Poland.

The study is designed to evaluate real-world practices related to the use of point-of-care lung ultrasound (LUS) in the decision-making process for surfactant therapy in neonates with Respiratory Distress Syndrome (RDS). The investigation is aligned with evolving European neonatal care guidelines that recommend incorporating LUS findings alongside traditional oxygen thresholds (FiO₂) when determining surfactant need.

All enrolled neonates will undergo a baseline lung ultrasound within the first 6 hours of life, prior to surfactant administration. LUS scoring will follow a validated 5-point scale (0-4) per lung quadrant, resulting in a total score between 0-16. A second LUS examination will be performed between 24 and 30 hours after surfactant administration to assess treatment response and identify any asymmetry in lung aeration, defined as a side-to-side LUS score difference ≥2 points.

In a subset of centers that routinely conduct neonatal hemodynamic assessments, echocardiographic evaluation of the main pulmonary artery (MPA) and ascending aorta (AA) diameters will be carried out. The MPA-to-AA ratio will serve as a surrogate marker of pulmonary vascular resistance and potential pulmonary hypertension. A ratio >1.3 will be considered indicative of clinically significant pulmonary arterial hypertension, consistent with published literature.

The surfactant treatment (product: Curosurf) will be administered per standard clinical practice, including both LISA (Less Invasive Surfactant Administration) and INSURE (INtubation, SURfactant administration, Extubation) methods. The mode of surfactant delivery and timing of administration will be recorded, as will any need for redosing.

Comprehensive clinical data-including gestational age, birth history, comorbidities, oxygenation parameters (SpO₂/FiO₂), and level and duration of respiratory support-will be collected through the neonatal hospital stay. Respiratory support will be categorized into escalating classes from spontaneous breathing to mechanical ventilation, to allow stratified analysis of post-surfactant respiratory outcomes.

The study will also explore associations between post-treatment lung ultrasound asymmetry, mode of surfactant delivery, and the presence of pulmonary comorbidities using multivariable logistic regression modeling.

All data will be collected in accordance with good clinical practice and applicable data protection regulations. As a non-interventional study, ULISSES is intended to provide evidence on the integration of bedside imaging into neonatal care, without altering routine clinical management.

The planned study duration is from end-July 2025 to December 2026.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates (gestational age <37 weeks) with established Respiratory Distress Syndrome (RDS) or at risk for RDS
* Decision of the use of surfactant by the attending physician

Exclusion Criteria:

* Presence of major congenital abnormalities of the respiratory system
* Infants requiring primary intubation and mechanical ventilation in the delivery room

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes preterm neonates born before 37 weeks of gestation with diagnosed or suspected Respiratory Distress Syndrome (RDS) who are considered for surfactant (SF) therapy based on the attending physician's judgment. Only infants managed initially without delivery room intubation are eligible, ensuring a baseline lung ultrasound (LUS) can be performed before SF administration.
  Participants will be recruited from tertiary neonatal intensive care units in Poland, all experienced in neonatal ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adoption of lung ultrasound in treatment decisions | 1st day of life
  The rate of surfactant treatment decisions based on lung ultrasound score (LUS)* versus those based on oxygen requirement**.
  *Definition of LUS-guided treatment: LUS score ≥6 points and FiO2 ≤0.30 before surfactant administration;
  **Definition of FiO2-guided treatment:: FiO2 >0.30, regardless of LUS score value before surfactant administration.

SECONDARY OUTCOMES:
Lung aeration asymmetry | From the time of SF administration to 24 hours (±6 hours) after the dose
  Percentage of infants presenting with the side-to-side lung ultrasound score difference ≥2 points at 24 hours after surfactant (SF) administration

OTHER OUTCOMES:
Vascular resistance in the pulmonary circulation. | From the time of SF administration to 24 hours (±6 hours) after the dose
  Changes in the Main Pulmonary Artery to Ascending Aorta ratio (MPA-to-AA) at 24 hours post-surfactant (SF) compared to pre-SF value

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Neonatology, Czerwiakowski Hospital at Siemiradzki st., Cracow, Poland, Krakow
  - Department of Neonatology and Neonatal Intensive Care, Medical University of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No
In accordance with the data protection policies of the Principal Investigator's institution, individual participant data (IPD) cannot be shared with external researchers